CLINICAL TRIAL: NCT06855953
Title: Vitamin K Supplementation to Improve Cognition of Patients With Coronary Heart Disease: a Randomized Controlled Pilot Study
Brief Title: Vitamin K and Cognition in Coronary Heart Disease (NutriCog)
Acronym: Nutricog
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2022-3025; (FRN) 183781_1 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2025-02-20; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease (CHD); Cognition; Cerebral vasoreactivity; Nutrition; Heart disease; Cardiovascular disease; Vitamins; Micronutrients; Vitamin K; Vitamin K1
MeSH Terms: conditions — Coronary Disease; Heart Diseases; Cardiovascular Diseases | interventions — Vitamin K

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement: Vitamin K (Experimental): Participants receive 0.5 mg/day phylloquinone orally for 12 weeks
  Interventions: Dietary Supplement: Vitamin K
- Dietary Supplement: Placebo (Placebo Comparator): Participants receive daily placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K — Participants receive 0.5 mg/day phylloquinone orally for 12 weeks
  Arms: Dietary Supplement: Vitamin K
Dietary Supplement: Placebo — Participants receive daily placebo for 12 weeks
  Arms: Dietary Supplement: Placebo

SUMMARY:
The purpose of this pilot study is to obtain a preliminary assessment of the effect of VK supplementation on cognitive performance and vascular function in adults with stable Coronary Heart Disease (CHD)

DETAILED DESCRIPTION:
The overall goal of this study is to obtain a preliminary assessment of the effect of a VK1 (phylloquinone) supplementation on cognitive performance (primary outcome) and vascular function (secondary outcome) in adults with stable CHD. Specifically, the investigators will conduct a double-blind, 2-armed, parallel-group intervention study in which 40 men and women aged 60 years and over with stable CHD will be randomly assigned to 0.5 mg phylloquinone per day or matching placebo for a period of 3 months. All participants will have signed a written consent form before taking part in the study

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 60 years and older
* Medically documented stable Coronary Heart Disease (CHD)
* Daily dietary intakes of phylloquinone <150 mcg
* Non-consumption of vitamin K supplements (i.e. K1 or K2, singly or in combination with other nutrients), or other cognitive aids
* Good French or English understanding
* Physical exercise not exceeding 2.5 hours/week of moderate to vigorous aerobic activity
* Capacity and willingness to sign informed consent

Exclusion Criteria:

* Recent acute coronary syndrome (<3 months) or recent coronary revascularization (bypass surgery or percutaneous coronary intervention, <3 months)
* Known left ventricular dysfunction (LVEF < 40%) or chronic heart failure
* Recent modification of medication (<2 weeks)
* Warfarin (Coumadin) use
* Cognitive impairment (based on telephone version of the Mini-Mental State Examination test, score <19/23)
* Diagnosis of depression or uncontrolled anxiety
* Malabsorption disorder (advanced liver disease, Crohn's disease)
* Patient with auditory or vision impairments not properly corrected by glasses or hearing aids
* Unable to read the informed consent form or unable to understand the oral explanations provided by the assessor

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in general cognitive functioning | Baseline and post-intervention at 12 weeks
  Montreal Cognitive Assessment (0-30 score, with a higher score indicating a better cognitive functioning)
Change in processing speed | Baseline and post-intervention at 12 weeks
  Processing speed is assessed using the Coding subtest from the Wechsler Adult Intelligence Scale (WAIS)IV. The participant is asked to reproduce, as rapidly as possible, a series of symbols associated with digits in a 2-min time period
Change in executive functions | Baseline and post-intervention at 12 weeks
  Executive function is assessed using
  1. Delis-Kaplan Executive Function System (D-KEFS) subtests [Trail Making Test; Phonological and Semantic Fluency test [Letters P, T, L (60s maximum); Categories: animals, men's names (60s maximum)]
  2. WAISIV subtests ("Switching" between naming fruit and furniture (60s maximum)]
  3. Neuropeak platform developed by Dr Bherer's laboratory: dual-task (divided attention) and n-back (working memory and updating). These tasks are tablet/computer-based
  As these tests use different scales, z-scores will be calculated for the different tests and a composite z-score will be generated for the domain
Change in episodic memory | Baseline and post-intervention at 12 weeks
  Episodic memory is assessed using:
  1. Rey auditory verbal learning test (RAVLT). Score 0-75, with a higher score indicating a better memory
  2. Digit span, a test that requires participants to repeat series of digits of increasing length
  As these tests use different scales, z-scores will be calculated for the different tests and a composite z-score will be generated for the domain

SECONDARY OUTCOMES:
Change in cerebral autoregulation - middle cerebral arteries | Baseline and post-intervention at 12 weeks
  Variations of cerebral blood flow velocity at the level of the middle cerebral artery will be measured in response to hypercapnic breathing using transcranial Doppler (TCD)
Change in cerebral pulsatility - middle cerebral arteries | Baseline and post-intervention at 12 weeks
  Pulsatility will be measured as the normalized difference of relative blood flow velocities between systole and diastole, using TCD in the middle cerebral arteries
Change in peripheral endothelial function | Baseline and post-intervention at 12 weeks
  Brachial artery flow-mediated dilation (FMD) will be quantified noninvasively by measuring blood velocity in the brachial artery and its diameter before and after 5 minutes of forearm hypoxia, using a high-resolution ultrasound device
Central arterial stiffness | Baseline and post-intervention at 12 weeks
  Central arterial stiffness will be assessed by measuring the carotid-femoral pulse-wave velocity (cfPWV), using a non-invasive surface tonometer

CONTACTS AND LOCATIONS:
Overall Officials: Guylaine Ferland, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published
Supporting Information: Study Protocol
Time Frame: Study protocol will be submitted for publication once the study registration process is completed